CLINICAL TRIAL: NCT06131580
Title: Continuation of an Open-label, Multi-center Study to Assess Long Term Safety in Canadian Patients With Endogenous Cushing's Syndrome Who Have Completed Prior Recordati-sponsored Osilodrostat (LCI699) Study LCI699C2X01B and Are Judged by the Investigator to Benefit From Continued Treatment With Osilodrostat
Brief Title: Canadian Continuation of Roll-over Study in Patients With Endogenous Cushing's Syndrome
Acronym: ISS-CA-2023
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: RECORDATI GROUP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MP-02-2024-11788; 278454 (Other: Health Canada)
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-10

CONDITIONS: Endogenous Cushing Syndrome
Keywords: Endogenous Cushing syndrome; Cushing syndrome; osilodrostat; long term safety; Canada
MeSH Terms: conditions — Cushing Syndrome | interventions — Methods; Therapeutics

STUDY DESIGN:
Intervention Model Description: This is a multi-center (four sites in Canada), open-label study to evaluate the long term safety of osilodrostat in 7 patients currently being treated in a Global Recordati-sponsored study (LCI699C2X01B) and who are judged by their doctor as benefiting from the current study treatment. The study is expected to remain open for approximately 2 years from EOT (end of trial) visit for each patient in roll-over study. Patients will continue to be treated in this study until they are no longer benefiting from their osilodrostat treatment as judged by the Investigator, until one of the protocoldefined discontinuation criteria is met. Additionally, Company (RRD) agrees to provide osilodrostat for investigational use through the study until patients can transition to commercially available and reimbursed drug in patients' province, as long as there is a path, as determine by RRD Canada Inc., to reimbursement.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participant Group/Arm (Other): Other: osilodrostat
  open label, with patients receiving same dose as provided in the parent study
  Interventions: Drug: Intervention/Treatment

INTERVENTIONS:
Drug: Intervention/Treatment — Drug: osilodrostat
  - osilodrostat, in the form of film coated tablets for oral administration, in the following tablet strengths: 1mg, 5mg, 10mg. Each strength has unique tablet size, colour and imprint.

SUMMARY:
The purpose of this study is to continue the evaluation of long-term safety of osilodrostat in 7 Canadian patients who have already received osilodrostat treatment in a previous Global Recordati-sponsored roll-over study and who, based on investigators' judgement, will continue benefiting with its administration.

DETAILED DESCRIPTION:
There will be no screening period for this study. Eligible subjects can start their treatment with osilodrostat as soon as they are enrolled in the study. The first study visit will be scheduled at the time of the last study visit for the parent study. Subjects must return to the study center at least on a quarterly basis (every 12 weeks ± 2 weeks) for safety and clinical benefit assessments, and resupply of study medication. Drug dispensing and administration information and adverse events will be collected. The subject may return to the clinic at any given time as per standard of care or treating physician recommendation; however, only the quarterly study visits will be recorded in the Case Report Form (CRF). Study medication dispensed will be recorded in the CRF dose administration page.

All adverse events and serious adverse events, including pregnancy, will be collected throughout the study. Subjects will continue to be treated in this roll-over study until they are no longer benefiting from their osilodrostat treatment as judged by the Investigator or until osilodrostat is commercially available or until one of other discontinuation criteria is met.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is currently participating in a Global Recordati-sponsored roll-over study receiving osilodrostat for any type of endogenous CS and has fulfilled all their requirements in the parent study.
2. The patient is currently benefiting from treatment with osilodrostat, as determined by the Investigator.
3. Patient has demonstrated compliance, as assessed by the Investigator, with the parent roll-over study protocol requirements.
4. Willingness and ability to comply with scheduled visits and treatment plans.
5. Written informed consent obtained prior to enrolling into the study

Exclusion Criteria:

1. Patient has been permanently discontinued from osilodrostat study treatment in the parent roll-over Recordati-sponsored study.
2. New patients not previously enrolled in parent roll-over Recordatisponsored study.
3. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory evaluation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2023-10-24 (Actual); Primary Completion 2025-11-24 (Estimated); Study Completion 2025-11-24 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse/serious adverse events | up to 2 years
  To evaluate long term safety

SECONDARY OUTCOMES:
Percentage of patients with clinical benefit | up to 2 years
  clinical benefit as assessed by the investigator

CONTACTS AND LOCATIONS:
Overall Officials: André Lacroix, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (3):
- Canada (3):
  - University of Alberta Hospital - Alberta Diabetes Institute, Edmonton, Alberta
  - Nova Scotia Health, Halifax, Nova Scotia
  - CHUS Sherbrooke, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No